CLINICAL TRIAL: NCT05573581
Title: Effect of Botox Injection in Anterior Belly of Digastric on Skeletal Relapse Following Mandibular Advancement Surgery (Randomized Controlled Trial)
Brief Title: Effect of Botox Injection in Anterior Belly of Digastric on Skeletal Relapse Following Mandibular Advancement Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, aya abd el rhman abd el atty, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01147686914
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Orthognathic Relapse
Keywords: mandibular advancement; orthognathic relapse
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox injection group (Experimental): Botox injection in anterior belly of digastric before mandibular advancement orthognathic surgery
  Interventions: Drug: Botox
- placebo group (No Intervention): no injection before surgery

INTERVENTIONS:
Drug: Botox — Botulinum toxin type A will be first injected into anterior belly of digastric muscles 2-3 days prior to any surgical intervention (for the BTX to be clinically effective)(Sadick and Matarasso 2004). A total of 20 U of Botox will be injected bilaterally by using 25g needle, 1 cc insulin syringe through extraoral approach in 4 point
  Other Names: botulinum toxin type A
  Arms: Botox injection group

SUMMARY:
The purpose of this study is to test whether Botox injection in anterior belly of digastric muscle in BSSO for mandibular advancement surgery could reduce the tendency of postoperative relapse.

Research question:

(P) In patient has skeletal class II mandibular retrognathism, (I) will Botox injection in anterior belly of digastric. (O) Affect the relapse of the mandible after mandibular advancement orthognathic surgery?

Participants will be undergo Botox injection in anterior belly of digastric and bilateral sagittal split surgery

DETAILED DESCRIPTION:
In the intervention group:

Botulinum toxin type A will be first injected into anterior belly of digastric muscles 2-3 days prior to any surgical intervention (for the BTX to be clinically effective). A total of 20 U of Botox will be injected bilaterally by using 25g needle, 1 cc insulin syringe through extra oral approach in 4 point.

Intra-operative procedures:

Access through a vestibular Sagittal split incision for mandible will be carried out. Dissection and reflection to reach the bone will be carried out.

* The cutting guide of the mandible will be placed onto the exposed bony surface and manipulated to the best fit. Then, the guide will be fixed using four 2.0-mm screws to avoid any mobilization during drilling of the reference holes. Sixteen reference holes will be established using the cutting guide; eight on each side.
* Then, a reciprocating saw will be used to perform the planned bilateral sagittal split osteotomy. After adequate mandibular mobilization and removal of bony interferences, the mandible will be repositioned using the patient-specific osteosynthesis material guided by the previously established reference holes and fixed using 2.0-mm screws.
* In Bi-max surgery the maxillary cutting guide will be fixed in the same manner and Lefort I osteotomy will be carried out.
* After adequate mobilization, the maxilla will be repositioned by the patient specific osteosynthesis material using the reference holes made by cutting guide and fixed using 2.0-mm screws.
* All incisions were closed with 4-0 resorbable sutures.

ELIGIBILITY:
Inclusion Criteria:

* Patients need bilateral sagittal split osteotomy for correction of skeletal class II malocclusion (mandibular retrognathism).
* Age of the patient above 18 years.
* All patients are free from any systemic disease that may affect normal bone healing.

Exclusion Criteria:

* Patient with history of facial bone trauma, cleft lip or palate.
* Intra-bony lesions or infections that may interfere with surgery.
* Previous orthognathic surgeries.
* Patients with relative contraindications to (BTX) injection such as pregnancy, lactation, neuromuscular diseases (e.g., myasthenia gravis), motor neuron disease, allergy to any of the components of (BTX).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
relapse | 6 month
  relapse in mandibular advancement